CLINICAL TRIAL: NCT06743100
Title: An Expanded Access Program for the Non-invasive Characterization of Glioma or Treatment Related Change Utilizing Fluorine (F-18) Floretyrosine (18F-FET, TLX101-CDx)
Brief Title: 18F-Floretyrosine Expanded Access Program
Status: Available | Type: Expanded Access
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 18F-TLX101-CDX-002
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Glioma (Any Grade) in the Brain
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Diagnostic Test: 18F-Floretyrosine — Single IV administration on Day 0, followed by a PET/CT or PET/MR diagnostic scan 20-40 minutes after the IV administration of 18F-Floretyrosine.

SUMMARY:
The aim of this Expanded Access Program (EAP) is to enable the use of 18F-Floretyrosine with positron emission tomography/computed tomography (PET/CT) or positron emission tomography/magnetic resonance (PET/MR) imaging to noninvasively detect tumor burden or treatment related change to assist in optimal management of patients with glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Written and voluntarily given informed consent. Pediatric patients (<18 years of age) will provide assent along with parental/legal guardian /caregiver consent according to IRB requirements.
2. Male or female ≥ 3 years of age at time of consent/assent
3. Diagnosis or clinical suspicion of glioma (any grade) in the brain
4. At the time of screening have undergone therapy for glioma
5. Indeterminate MR findings for disease recurrence or progression versus treatment related changes (pseudoprogression or pseudoresponse) requiring further diagnostic procedures within 60 days prior to the 18F-Floretyrosine PET imaging
6. Willing and able to lie still for at least 40 minutes in an enclosed space for the imaging procedure, or if medically necessary, able to tolerate standard institutions procedures for sedation and/or anesthesia.

Exclusion Criteria:

1. Participant cannot be safely scanned due to devices, implants, foreign and/or metallic objects in or on the body that are not MR compatible, unless a clinical judgement is made that the participant's diagnostic needs can instead be met by diversion to 18F-Floretyrosine imaging by PET/CT (making the magnetic field compatibility an irrelevant safety concern).
2. Women who are pregnant or breastfeeding.
3. Women of childbearing potential who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for the duration of the program (Day 0 to Day 2).
4. Serious non-malignant disease (e.g., psychiatric, infectious, autoimmune, or metabolic), that may interfere with the objectives of the program or with the safety or compliance of the participant, as judged by the Investigator.
5. Mental impairment that may compromise the ability to give informed consent/assent and comply with the requirements of the program as judged by the Investigator.
6. Exposure to any experimental diagnostic or therapeutic drug within 30 days from the date planned administration of 18F-Floretyrosine.
7. Known hypersensitivity to floretyrosine or tyrosine derivatives.
8. Unable to tolerate the program procedures.

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - CU Anschutz / University of Colorado, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Baltimore, Baltimore, Maryland
  - Kettering Health Main Campus, Kettering, Ohio
  - University Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University Wisconsin Madison, Madison, Wisconsin